CLINICAL TRIAL: NCT05676320
Title: A Multicentre, Single-blind, RCT to Document the Safety and Efficacy of the Use of a Bone Cement With or Without Inossia® Cement Softener for Patients With Vertebral Compression Fractures
Brief Title: Investigating Bone Cement With or Without Inossia® Cement Softener for Vertebral Compression Fractures
Acronym: SOFTBONE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inossia AB (Industry)
Collaborators: EIT Health (Other); Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SOFTBONE 1512:1
Record Dates: First submitted 2022-12-14; First posted 2023-01-09 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Vertebral Compression Fracture
Keywords: vertebral compression fracture; bone cement; vertebroplasty; kyphoplasty; osteoporosis; softener
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- V-Flex (Experimental): Bone cement including Inossia® Cement Softener
  Interventions: Device: V-Flex
- V-Steady (Active Comparator): Bone Cement alone
  Interventions: Device: V-Steady

INTERVENTIONS:
Device: V-Flex — Bone cement including Inossia® Cement Softener. Treatment for vertebral compression fracture
  Arms: V-Flex
Device: V-Steady — Bone Cement alone
  Arms: V-Steady

SUMMARY:
The overall purpose of conducting this study is to evaluate the safety and efficacy of V-Flex and V-Steady for augmentation of osteoporotic vertebral compression fractures and to verify that adding a cement softener into a PMMA bone cement is comparable to a PMMA bone cement alone (V-Steady).

DETAILED DESCRIPTION:
The clinical investigation is a prospective, single-blind, controlled multi-center study of vertebral compression fractures treated by vertebroplasty or kyphoplasty with PMMA alone (V-Steady) or PMMA mixed with Inossia® Cement Softener (V-Flex).

The overall purpose of conducting this study is to confirm the safety and efficacy of Inossia® Cement Softener mixed with PMMA for augmentation of osteoporotic vertebral compression fractures and to verify that the V-Flex is, at least, comparable (non-inferior) to the PMMA products used today.

All eligible patients will be invited to participate in the study. A total of 150 patients will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any study-related activities (study-related activities are any procedures that would not have been performed during normal management of the patient, i.e. standard of care);
* Symptomatic osteoporotic vertebral compression fracture without prior or not responding to medical treatment within 6 months;
* Maximum of 1 level of vertebral compression fractures eligible for treatment localized at level Th5 to L5 and verified by MRI or bone scan;
* Height reduction of the affected vertebra(e) with an anterior wall compression of not exceeding 60% compared to the nearest normal vertebral body determined by X-ray;
* Have pain correlating to the fractured levels requiring regular analgesic intake and/or causing substantial disability of daily life;
* Pain score ≥ 40 mm measured by VAS correlating to at least one of the fracture levels (scale 0 - 100 mm) at the screening visit;
* Oswestry Disability Index > 20 (0 - 100 scale);
* SF-12PCS Index < 80 (0 - 100 scale);
* Patient with a communicative ability to understand the procedure and participate in the study and comply with the follow up program.

Exclusion Criteria:

* Patients below 18 years;
* Any burst fracture;
* Unstable fractures defined by neurological deficit or interspinous process widening as evaluated by the Investigator, as well as kyphosis > 30°, translation > 4 mm;
* Established or suspected malignancy of the fractured vertebra. Hemangioma of the fractured vertebra;
* High energy trauma or clinical diagnosis of herniated nucleus pulposus or severe spinal stenosis as suggested by progressive weakness;
* Have neurologic symptoms or deficits, or radiculopathy related to the fractured vertebrae;
* Patients with extremely high BMI, i.e. BMI ≥ 40;
* Previously treated with vertebroplasty or kyphoplasty;
* Patients with concomitant diseases which may be worsened by invasive treatment of the fracture such as e.g. severe cardiopulmonary dysfunction (including aortic aneurysm), as judged by the Investigator
* Irreversible coagulopathy or bleeding disorder. Note regarding reversible coagulopathies: Patients on Coumadin or other anticoagulants may participate. Investigators should follow routine practices for perioperative discontinuation and re- initiation of anticoagulants;
* Active systemic infection or local skin infection at the puncture site;
* Pregnancy or breast-feeding;
* Patients with known chemical dependency or drugs or with a medical history of drug abuse;
* Patients who are serving prison sentence;
* Have participated in another investigational study within 30 days prior to inclusion
* Pacemaker
* Previous or active radiotherapy affecting the spine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2021-03-11 (Actual); Primary Completion 2025-10-20 (Actual); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
New fractures | 1 year
  To assess the effectiveness after administration of V-Flex compared to V-Steady as measured by reduction of new radiologically confirmed fractures.
Location of fractures | 1 year
  Assess the location of new fractures: adjacent or non-adjacent to the treated vertebral or re-fractures of the treated vertebra after administration of the investigational device compared to PMMA.
Timing of fractures | 1 year
  Assess the timing of adjacent, non-adjacent and re-fractures of the treated vertebra after administration of the investigational device compared to PMMA.

SECONDARY OUTCOMES:
Function by ODI | 24 months
  Assess the change in function at time points 5 days, 3 months, 12 months, and 24 months after administration of the investigational device compared to PMMA as measured by Oswestry Disability Index (ODI): scale 0-100% where a higher score means a worse outcome
Pain measured by VAS | 24 months
  Assess the change in back pain at time points 5 days, 3 months, 12 months, and 24 months after administration of the investigational device compared to PMMA as measured by Visual Analogue Scale (VAS): scale 0-100, where 0 is no pain and 100 is the worst pain imaginable
Health related quality of life by SF-12 | 24 months
  Assess the change in health related quality of life at time points 5 days, 3 months, 12 months, and 24 months after administration of the investigational device compared to PMMA as measured by SF-12: scale 0-100 where a higher score means a better outcome
Safety measured by adverse events | 24 months
  Asses the safety of Inossia™ Cement Softener as measured by adverse events
Hospital Beds | 1 week
  Record the number of hospital bed days (within hospital, nursing home, etc.) during the first week
The vertebral height | 24 month
  The vertebral height at 12 months and 24 months compared to baseline by X-ray (Average Mid Vertebral Body Height)
Analgesic use | 24 months
  Record the analgesic use at time points 5 days, 3 months, 12 months, and 24 months after administration of the investigational device compared to PMMA and compare to the WHO analgestic ladder
Osteoporotic treatment regimen checklist | 24 months
  Record the osteoporotic treatment regimen at time points 5 days, 3 months, 12 months, and 24 months after administration of the investigational device compared to PMMA

CONTACTS AND LOCATIONS:
Overall Officials: David Noriega, Principal Investigator — University Hospital in Valladolid
Locations (7):
- Beam Radiology, Calgary, Alberta, Canada
- Germany (2):
  - Mannheim University Hospital, Mannheim
  - Hospital in Mechernich, Mechernich
- Lodz University Hospital, Lodz, Poland
- Spain (3):
  - Clínico San Carlos, Madrid
  - Puerta de Hierro, Madrid
  - University Hospital in Valladolid, Valladolid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooper C, Atkinson EJ, O'Fallon WM, Melton LJ 3rd. Incidence of clinically diagnosed vertebral fractures: a population-based study in Rochester, Minnesota, 1985-1989. J Bone Miner Res. 1992 Feb;7(2):221-7. doi: 10.1002/jbmr.5650070214. PMID 1570766
- [Background] Leidig G, Minne HW, Sauer P, Wuster C, Wuster J, Lojen M, Raue F, Ziegler R. A study of complaints and their relation to vertebral destruction in patients with osteoporosis. Bone Miner. 1990 Mar;8(3):217-29. doi: 10.1016/0169-6009(90)90107-q. PMID 2322694
- [Background] International Committee of Medical Journal Editors. Uniform requirements for manuscripts submitted to biomedical journals. N Engl J Med. 1997 Jan 23;336(4):309-15. doi: 10.1056/NEJM199701233360422. No abstract available. PMID 8995096
- [Background] International Conference on Harmonisation. ICH Harmonised Tripartite Guideline. Good Clinical Practice. 1-5-1996.
- [Background] Code of Federal Regulations. Title 21, Volume 8. Part 812, Investigational Device Exemptions, Revised 2006.
- [Background] World Medical Association. Declaration of Helsinki. Ethical Principles for Medical Research Involving Human Subjects. 52nd WMA General Assembly, Edinburgh, Scotland, October 2000. Last amended with Note of Clarification of Paragraph 29 by the WMA General Assembly, Washington 2002 and Note of Clarification on Paragraph 30 by the WMA General assembly, Tokyo 2004.
- [Background] de Bruin TW. Iodide-induced hyperthyroidism with computed tomography contrast fluids. Lancet. 1994 May 7;343(8906):1160-1. doi: 10.1016/s0140-6736(94)90265-8. No abstract available. PMID 7910248
- [Background] ICH Harmonised Tripartite Guideline. Statistical principles for clinical trials. International Conference on Harmonisation E9 Expert Working Group. Stat Med. 1999 Aug 15;18(15):1905-42. No abstract available. PMID 10532877
- [Background] Lane JI, Maus TP, Wald JT, Thielen KR, Bobra S, Luetmer PH. Intravertebral clefts opacified during vertebroplasty: pathogenesis, technical implications, and prognostic significance. AJNR Am J Neuroradiol. 2002 Nov-Dec;23(10):1642-6. PMID 12427615
- [Background] Trout AT, Kallmes DF, Gray LA, Goodnature BA, Everson SL, Comstock BA, Jarvik JG. Evaluation of vertebroplasty with a validated outcome measure: the Roland-Morris Disability Questionnaire. AJNR Am J Neuroradiol. 2005 Nov-Dec;26(10):2652-7. PMID 16286418
- [Background] Trout AT, Gray LA, Kallmes DF. Vertebroplasty in the inpatient population. AJNR Am J Neuroradiol. 2005 Aug;26(7):1629-33. PMID 16091505
- [Background] Layton KF, Thielen KR, Koch CA, Luetmer PH, Lane JI, Wald JT, Kallmes DF. Vertebroplasty, first 1000 levels of a single center: evaluation of the outcomes and complications. AJNR Am J Neuroradiol. 2007 Apr;28(4):683-9. PMID 17416821
- [Background] Voormolen MH, van Rooij WJ, Sluzewski M, van der Graaf Y, Lampmann LE, Lohle PN, Juttmann JR. Pain response in the first trimester after percutaneous vertebroplasty in patients with osteoporotic vertebral compression fractures with or without bone marrow edema. AJNR Am J Neuroradiol. 2006 Aug;27(7):1579-85. PMID 16908585
- [Background] Palussiere J, Berge J, Gangi A, Cotten A, Pasco A, Bertagnoli R, Jaksche H, Carpeggiani P, Deramond H. Clinical results of an open prospective study of a bis-GMA composite in percutaneous vertebral augmentation. Eur Spine J. 2005 Dec;14(10):982-91. doi: 10.1007/s00586-003-0664-2. Epub 2005 Jun 2. PMID 15931511
- [Background] Cortet B, Cotten A, Boutry N, Flipo RM, Duquesnoy B, Chastanet P, Delcambre B. Percutaneous vertebroplasty in the treatment of osteoporotic vertebral compression fractures: an open prospective study. J Rheumatol. 1999 Oct;26(10):2222-8. PMID 10529144
- [Background] Prather H, Van Dillen L, Metzler JP, Riew KD, Gilula LA. Prospective measurement of function and pain in patients with non-neoplastic compression fractures treated with vertebroplasty. J Bone Joint Surg Am. 2006 Feb;88(2):334-41. doi: 10.2106/JBJS.D.02670. PMID 16452745
- [Background] Vogl TJ, Proschek D, Schwarz W, Mack M, Hochmuth K. CT-guided percutaneous vertebroplasty in the therapy of vertebral compression fractures. Eur Radiol. 2006 Apr;16(4):797-803. doi: 10.1007/s00330-005-0021-4. Epub 2005 Dec 7. PMID 16333624
- [Background] Gaughen JR Jr, Jensen ME, Schweickert PA, Kaufmann TJ, Marx WF, Kallmes DF. Lack of preoperative spinous process tenderness does not affect clinical success of percutaneous vertebroplasty. J Vasc Interv Radiol. 2002 Nov;13(11):1135-8. doi: 10.1016/s1051-0443(07)61955-1. PMID 12427813
- [Background] Do HM, Kim BS, Marcellus ML, Curtis L, Marks MP. Prospective analysis of clinical outcomes after percutaneous vertebroplasty for painful osteoporotic vertebral body fractures. AJNR Am J Neuroradiol. 2005 Aug;26(7):1623-8. PMID 16091504
- [Background] Fairbank JC, Pynsent PB. The Oswestry Disability Index. Spine (Phila Pa 1976). 2000 Nov 15;25(22):2940-52; discussion 2952. doi: 10.1097/00007632-200011150-00017. PMID 11074683
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Voormolen MH, Mali WP, Lohle PN, Fransen H, Lampmann LE, van der Graaf Y, Juttmann JR, Jansssens X, Verhaar HJ. Percutaneous vertebroplasty compared with optimal pain medication treatment: short-term clinical outcome of patients with subacute or chronic painful osteoporotic vertebral compression fractures. The VERTOS study. AJNR Am J Neuroradiol. 2007 Mar;28(3):555-60. PMID 17353335
- [Background] Guidance Document for the Preparation of IDEs for Spinal Systems, January 13, 2000.
- [Background] Clinical Trial Considerations:Vertebral Augmentation Devices to Treat Spinal lnsufficiency Fractures, October 24, 2004.
- [Background] Clauss W. How big is the risk of an examination with x-ray contrast media of patients with known hypersensitivity to CM and for allergic patients? In Dawson P and Clauss W (eds.): Contrast media in practice, 2nd edition, Springer-Verlag, Berlin-Heidelberg, 1999:98-99.
- [Background] Katayama H, Yamaguchi K, Kozuka T, Takashima T, Seez P, Matsuura K. Adverse reactions to ionic and nonionic contrast media. A report from the Japanese Committee on the Safety of Contrast Media. Radiology. 1990 Jun;175(3):621-8. doi: 10.1148/radiology.175.3.2343107.
- [Background] Wijn D and Mullen V. Biocompatibility of Acrylic lmplants. In Biocompatibility of Clinical lmplant Materials. Edited,CRC Press, 1981.
- [Background] Trout AT, Kallmes DF, Kaufmann TJ. New fractures after vertebroplasty: adjacent fractures occur significantly sooner. AJNR Am J Neuroradiol. 2006 Jan;27(1):217-23. PMID 16418388
- [Background] Uppin AA, Hirsch JA, Centenera LV, Pfiefer BA, Pazianos AG, Choi IS. Occurrence of new vertebral body fracture after percutaneous vertebroplasty in patients with osteoporosis. Radiology. 2003 Jan;226(1):119-24. doi: 10.1148/radiol.2261011911. PMID 12511679
- [Background] Grados F, Depriester C, Cayrolle G, Hardy N, Deramond H, Fardellone P. Long-term observations of vertebral osteoporotic fractures treated by percutaneous vertebroplasty. Rheumatology (Oxford). 2000 Dec;39(12):1410-4. doi: 10.1093/rheumatology/39.12.1410. PMID 11136886
- [Background] Kim CW, Minocha J, Wahl CE, Garfin SR. Response of fractured osteoporotic bone to polymethylacrylate after vertebroplasty: case report. Spine J. 2004 Nov-Dec;4(6):709-12. doi: 10.1016/j.spinee.2004.05.002. PMID 15597484
- [Background] McKiernan F, Faciszewski T, Jensen R. Quality of life following vertebroplasty. J Bone Joint Surg Am. 2004 Dec;86(12):2600-6. doi: 10.2106/00004623-200412000-00003. PMID 15590842
- [Background] Gill JB, Kuper M, Chin PC, Zhang Y, Schutt R Jr. Comparing pain reduction following kyphoplasty and vertebroplasty for osteoporotic vertebral compression fractures. Pain Physician. 2007 Jul;10(4):583-90. PMID 17660858
- [Background] Eck JC, Nachtigall D, Humphreys SC, Hodges SD. Comparison of vertebroplasty and balloon kyphoplasty for treatment of vertebral compression fractures: a meta-analysis of the literature. Spine J. 2008 May-Jun;8(3):488-97. doi: 10.1016/j.spinee.2007.04.004. Epub 2007 May 29. PMID 17588820
- [Background] Kado DM, Browner WS, Palermo L, Nevitt MC, Genant HK, Cummings SR. Vertebral fractures and mortality in older women: a prospective study. Study of Osteoporotic Fractures Research Group. Arch Intern Med. 1999 Jun 14;159(11):1215-20. doi: 10.1001/archinte.159.11.1215. PMID 10371229
- [Background] Cooper C, Atkinson EJ, Jacobsen SJ, O'Fallon WM, Melton LJ 3rd. Population-based study of survival after osteoporotic fractures. Am J Epidemiol. 1993 May 1;137(9):1001-5. doi: 10.1093/oxfordjournals.aje.a116756. PMID 8317445
- [Background] Silverman SL, Minshall ME, Shen W, Harper KD, Xie S; Health-Related Quality of Life Subgroup of the Multiple Outcomes of Raloxifene Evaluation Study. The relationship of health-related quality of life to prevalent and incident vertebral fractures in postmenopausal women with osteoporosis: results from the Multiple Outcomes of Raloxifene Evaluation Study. Arthritis Rheum. 2001 Nov;44(11):2611-9. doi: 10.1002/1529-0131(200111)44:113.0.co;2-n. PMID 11710717
- [Background] Nevitt MC, Ettinger B, Black DM, Stone K, Jamal SA, Ensrud K, Segal M, Genant HK, Cummings SR. The association of radiographically detected vertebral fractures with back pain and function: a prospective study. Ann Intern Med. 1998 May 15;128(10):793-800. doi: 10.7326/0003-4819-128-10-199805150-00001. PMID 9599190